CLINICAL TRIAL: NCT02861664
Title: A Study to Evaluate the Efficacy of an Experimental Occlusion Technology Dentifrice in the Relief of Dentinal Hypersensitivity
Brief Title: Assessment of the Efficacy of an Experimental Occlusion Technology Dentifrice in Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205794
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-06

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Test Dentifrice: Stannous fluoride (SnF2) (Experimental): Participants were instructed to apply a strip of dentifrice containing 0.454% stannous fluoride (SnF2) and 0.072% sodium fluoride (NaF) (1450 parts per million [ppm] fluoride in total) to cover the head of the toothbrush and brush their teeth for 1 timed minute, twice daily (morning and evening), following their normal routine. Participants were also permitted to rinse with tap water.
  Interventions: Other: Stannous fluoride (SnF2)
- Negative Control Dentifrice: Sodium monofluorophosphate (SMFP) (Active Comparator): Participants were instructed to apply a strip of dentifrice containing 1400ppm fluoride as sodium monofluorophosphate (SMFP) to cover the head of the toothbrush and brush their teeth for 1 timed minute, twice daily (morning and evening), following their normal routine. Participants were also permitted to rinse with tap water.
  Interventions: Other: Sodium monofluorophosphate (SMFP)

INTERVENTIONS:
Other: Stannous fluoride (SnF2) — Dentifrice containing 0.454% weight by weight (w/w) SnF2 and 0.072% w/w NaF
  Arms: Test Dentifrice: Stannous fluoride (SnF2)
Other: Sodium monofluorophosphate (SMFP) — Dentifrice containing 1400 ppm fluoride as SMFP
  Arms: Negative Control Dentifrice: Sodium monofluorophosphate (SMFP)

SUMMARY:
This study will evaluate the effectiveness of an experimental dentifrice containing stannous fluoride, an established dentine tubule occlusion technology, at reducing dentine hypersensitivity (DH) compared to a negative control dentifrice. The test and control dentifrices will be administered for a total of 8 weeks, with assessments (via evaporative air and tactile stimuli) at baseline, and after 4 and 8 weeks twice-daily use.

DETAILED DESCRIPTION:
This single centre, randomized, controlled, examiner-blind, 2 treatment arm, parallel group design study, stratified by maximum baseline Schiff sensitivity score (of the two selected teeth), with a treatment period of 8 weeks will investigate the clinical effectiveness of an experimental stannous fluoride dentifrice in the reduction of DH. DH will be assessed at Baseline, and after 4 and 8 weeks treatment to monitor clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Aged between 18 and 65 years inclusive
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon oral examination and absence of any condition that would impact on the participant's safety or well being or affect the individual's ability to understand and follow study procedures and requirements.
* At Screening-
* Self-reported history of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years.
* Good general oral health, with a minimum of 20 natural teeth.
* Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria; signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR), tooth with MGI score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1 and tooth with signs of sensitivity measured by qualifying evaporative air assessment (Schiff sensitivity score ≥1).
* At Baseline (Visit 2)-
* Minimum of two, non-adjacent accessible teeth (incisors, canines, premolars), that meet all of the following criteria i.e.
* Tooth with signs of sensitivity, measured by response to a qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff sensitivity score ≥ 2).

Exclusion Criteria

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit, previous participation in this study and participation in another tooth desensitizing treatment study within 8 weeks of the screening visit.
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes, presence of a condition which, in the opinion of the investigator is causing xerostomia.
* Dental prophylaxis within 4 weeks of Screening, tongue or lip piercing or presence of dental implants and gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Teeth bleaching within 8 weeks of Screening.
* Desensitising treatment within 8 weeks of screening (professional sensitivity treatments and non-dentifrice sensitivity treatments).
* Specific Dentition Exclusions For Test Teeth
* a) Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening
* b) Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* C) Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening (Participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients).
* Any subject who, in the judgment of the investigator, should not participate in the study, any condition which in the opinion of the investigator would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Daily doses of medication/treatments or traditional herbal ingredients/treatments which, in the opinion of the investigator, could interfere with the perception of pain (Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs and examples of herbal ingredients/treatments include clove oil, olive oil, or other treatments that are directly applied to the oral cavity for the treatment of oral health conditions).
* Currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline.
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Individuals who require antibiotic prophylaxis for dental procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wuhan, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in China.
Pre-assignment Details: A total of 273 participants were screened, out of which 135 participants were randomized to the study. 138 participants were not randomized because out of these, 135 participants did not meet the study criteria and 3 participants withdrew consent.
Period: Overall Study
Arm/Group | Test Dentifrice: Stannous Fluoride (SnF2) | Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP)
Started | 67 | 68
Completed | 67 | 67
Not Completed | 0 | 1
Not completed — Withdrawal of Consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the participants who were randomized, received at least one dose of the study treatment and provided at least one post-baseline assessment of efficacy.
Groups:
- Test Dentifrice: Stannous Fluoride (SnF2): Participants were instructed to apply a strip of dentifrice containing 0.454% SnF2 and 0.072% NaF (1450 ppm fluoride in total) to cover the head of the toothbrush and brush their teeth for 1 timed minute, twice daily (morning and evening), following their normal routine. Participants were also permitted to rinse with tap water.
- Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP): Participants were instructed to apply a strip of dentifrice containing 1400ppm fluoride SMFP to cover the head of the toothbrush and brush their teeth for 1 timed minute, twice daily (morning and evening), following their normal routine. Participants were also permitted to rinse with tap water.
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice: Stannous Fluoride (SnF2) | Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP) | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (8.21) | 41.9 (8.83) | 41.0 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 121
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 67 | 67 | 134
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Schiff Sensitivity Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The examiner assessed the participant's response to evaporative air stimulus, after the stimulation of each individual tooth, using the Schiff Sensitivity Scale as follows: 0 Participant does not respond to air stimulation, 1 Participant responds to air stimulus but does not request discontinuation of stimulus, 2 Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3 Participant responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicate improvement in sensitivity. Population: This baseline measurement was performed on ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy.
  score on a scale | 2.26 (0.393) | 2.23 (0.352) | 2.25 (0.372)
Tactile Threshold at Baseline [Mean (Standard Deviation); unit: gram (g)] — The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force has reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g. Population: This baseline measurement was performed on ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy.
  gram (g) | 11.1 (2.10) | 10.9 (2.29) | 11.0 (2.19)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 8
Description: The examiner assessed the participant's response to the evaporative air stimulus, after the stimulation of each individual tooth, using the Schiff Sensitivity Scale as follows: 0 Participant does not respond to air stimulation, 1 Participant responds to air stimulus but does not request discontinuation of stimulus, 2 Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3 Participant responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicate improvement in sensitivity.
Time Frame: At Baseline and Week 8
Population: ITT population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice: Stannous Fluoride (SnF2) | Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP)
Number analyzed (Participants) | 67 | 67
score on a scale | -0.94 (0.526) | -0.33 (0.699)
Statistical Analysis 1: Comparison: Test Dentifrice: Stannous Fluoride (SnF2) vs Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP); Test type: Other; p < .0001, ANCOVA — From ANCOVA model with change from baseline in Schiff Sensitivity Score as response and treatment and baseline Schiff sensitivity score as covariates; Least square (LS) mean difference = -0.6, 95% CI [-0.8 to -0.4] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favours first named dentifrice

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 4
Description: as for outcome 1
Time Frame: At Baseline and Week 4
Population: ITT population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy. Number of participants analyzed is number of participants from ITT population evaluated at Week 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice: Stannous Fluoride (SnF2) | Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP)
Number analyzed (Participants) | 66 | 67
score on a scale | -0.63 (0.570) | -0.10 (0.512)

3. Secondary Outcome: Change From Baseline in Tactile Threshold at Week 4 and 8
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force has reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g.
Time Frame: At Baseline, Week 4 and Week 8
Population: ITT population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy. Number of participants analyzed is the number of participants from ITT population evaluated at specific time point for each treatment arm respectively.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Test Dentifrice: Stannous Fluoride (SnF2) | Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP)
Number analyzed (Participants) | 67 | 67
g
  Change from baseline at Week 4: number analyzed (Participants) | 66 | 67
  Change from baseline at Week 4 | 4.8 (8.57) | 4.9 (12.31)
  Change from baseline at Week 8 | 10.4 (14.87) | 8.4 (16.73)

ADVERSE EVENTS:
Time Frame: Approximately 64 days
Groups:
- Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP): Participants were instructed to apply a strip of dentifrice containing 1400ppm fluoride as SMFP to cover the head of the toothbrush and brush with assigned dentifrice twice daily (morning and evening) for 1 timed minute. Participants were permitted to rinse with tap water.
Arm/Group | Test Dentifrice: Stannous Fluoride (SnF2) | Negative Control Dentifrice: Sodium Monofluorophosphate (SMFP)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68
Other Adverse Events (participants affected / at risk) | 0/67 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.